CLINICAL TRIAL: NCT01187121
Title: Evaluating A Drug Testing and Graduated Sanctions Program in Delaware
Acronym: DYT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Delaware (Other)
Collaborators: Delaware Department of Probation & Parole (Unknown)
Responsible Party: Daniel Joseph O'Connell, University of Delaware
Other Study IDs: 139855
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2010-08

CONDITIONS: Probationary Failure; Recidivism; Drug Relapse
Keywords: Graduated Sanctions; Probationary failure; recidivism; drug relapse; criminal justice
MeSH Terms: conditions — Recidivism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental: Those persons randomized to the Decide Your Time program.
- Standard Pracitice: Those persons randomized to the standard probationary practice condition.

SUMMARY:
The objective of this three year project funded by the National Institute of Justice is to conduct a program evaluation of the "Decide Your Time" program at the Hares Corner Office of the Delaware Department of Probation and Parole. The program is intended to provide an alternative to incarceration by monitoring chronic drug offenders through increased, regularly scheduled, known urinalysis testing, coupled with increasing sanctions and referral to treatment for positive tests. The program was designed and is being implemented by the Delaware Department of Probation and Parole. Offenders will become eligible for the program when they test positive for drugs at their initial probation intake at the Hare's Corner Probation Office in New Castle, Delaware or are moved from standard probation to intensive supervision due to failed urine tests. Due to budgetary constraints, the office lacks sufficient resources to place all eligible offenders into the program. The Department of Probation thus intends to randomly assign eligible offenders to either intensive supervision probation (ISP)(n=400) or the Decide Your Time program(n=400). Those in ISP will receive the normal intensive supervision requirements, including weekly visits and random urinalysis. Those in the enhanced condition will receive regularly scheduled urinalysis coupled with referral to treatment, if required, and a program of graduated sanctions. The Center for Drug and Alcohol Studies is conducting an evaluation of the program that involves examining data on effectiveness, and collecting and examining data on program implementation, and probation officer and client perspectives of how the program worked. It is hypothesized that those randomized to the Decide Your Time program will have fewer arrests, violations and positive urine screens upon program completion than those randomized to the control condition.

ELIGIBILITY:
Inclusion Criteria:

* sentenced to intensive supervision and fails a urine drug screen at the HAres Corner Probation office in Delaware

Exclusion Criteria:

* Clinical Diagnosis of DSM-IV Mental Illness
* Judge ordered Zero Tolerance program
* Sex Offender
* Less than sixty days on probation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Delaware Probationers who fail a urine screen are randomly assigned to either intensive supervision probation (ISP)(n=400) or the Decide Your Time program(n=400).
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2010-06

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J O'Connell, PhD, Principal Investigator — University of Delaware
Locations (1):
- New Castle Day Reporting Center at Hares Corner, 26 Parkway Circle, New Castle, Delaware, United States

REFERENCES:
- See also: Related Info — http://www.ojp.usdoj.gov/nij/topics/corrections/community/drug-offenders/decide-your-time.htm